CLINICAL TRIAL: NCT06906588
Title: Effects of Bilateral Upper Limb Robot-assisted Rehabilitation on Motor Recovery in Patients With Subacute Stroke: an Italian Multicenter Randomized Controlled Trial
Brief Title: Bilateral Robot-assisted Upper Extremity Rehabilitation on Motor Recovery in People With Subacute Stroke
Acronym: BILAX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele Roma (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 93/SR/24
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Stroke; Sabacute Stroke
Keywords: Upper limb rehabilitation; Bilateral Robot-Assisted Therapy-BRAT; stroke; subacute; Robotic rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: The study protocol will involve people diagnosed with stroke according to established inclusion and exclusion criteria who will be randomly assigned to one of the following groups:
  Experimental Group (EG) - robotic treatment for upper limb rehabilitation. Control group (CG) - conventional treatment for upper limb rehabilitation. The randomization will be carried out in a stratified way to have an even more homogeneous distribution in the two groups of subjects for the prognostic factors that play an important role in the treatment of people with stroke.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (EG) (Experimental): The experimental group (EG), in addition to the standard rehabilitation treatment, will perform one Bilateral Robot-Assisted Therapy-BRAT session per day through the Arm Light Exoskeleton Hybrid (Alex RS - Wearable Robotics) robotic system. Each participant will perform a total of 16+/-3 treatment sessions. The device that will be used have the CE (European Conformity) marking.
  Interventions: Device: Experimental
- Control Group (CG) (Active Comparator): The control group (CG), in addition to the standard routine rehabilitation treatment, will follow 45 minutes of conventional rehabilitation of the upper limbs without the use of technological devices. Each participant will perform a total of 16+/-3 conventional upper limb treatment sessions. The motor exercises will concern the rehabilitation of the upper limb and will be performed with a therapist who will personalize the treatment based on the clinical characteristics and needs of the patient.
  Interventions: Other: Control

INTERVENTIONS:
Device: Experimental — The experimental group (EG), in addition to the standard rehabilitation treatment, will perform one upper limb BRAT session per day through the Arm Light Exoskeleton Hybrid (Alex RS - Wearable Robotics) robotic system.. Each participant will perform a total of 16+/-3 treatment sessions with a frequency of 4 times a week for 4 consecutive weeks. During the first session, the device should be adjusted according to the patient's bilateral size and suspension angle. The selection of personalized exercises will be based on each patient's motor skills and the difficulty can be gradually increased during the treatment period. These modalities are shown to the patient with visual and motor feedback (force feedback). The duration of the single rehabilitation treatment is 45 minutes, of which 5 minutes are used for setting up the device, 10 minutes for assembly/disassembly, 10 minutes for unilateral treatment with the affected upper limb and 20 minutes for bilateral treatment.
  Arms: Experimental Group (EG)
Other: Control — The control group (GC), in addition to the standard routine rehabilitation treatment, will follow 45 minutes of conventional rehabilitation of the upper limbs without the use of technological devices. Each participant will perform a total of 16+/-3 conventional upper limb treatment sessions with a frequency of 4 times a week for 4 weeks. The motor exercises will concern the rehabilitation of the upper limb and will be performed with a therapist who will personalize the treatment based on the clinical characteristics and needs of the patient. Specifically, the treatment of the upper limb will be characterized by motor exercises (shoulder, elbow, wrist and hand), coordination and manual dexterity. Each session will consist of passive, active-assisted and active exercises.
  Arms: Control Group (CG)

SUMMARY:
The goal of this clinical trial is to study the clinical effects of a robotic rehabilitation treatment through a bilateral exoskeleton (Bilateral Robot-Assisted Therapy-BRAT) during standard rehabilitation, on motor recovery, compared to conventional arm re-education in people suffering from stroke in the subacute phase. The main question it aims to answer is what the effectiveness of Bilateral Robot-Assisted Therapy (BRAT) is in rehabilitating the upper limb in individuals with subacute stroke compared to conventional rehabilitation treatment in terms of motor function improvement as measured by the Fugl-Meyer Assessment - Upper Limb (FMA-UL), motor domain. Researchers will compare two groups (Experimental Group - EG and Control Group - CG) to see if the BRAT is more effective than conventional rehabilitation treatment in terms of motor recovery. Participants will be randomly assigned to one of the two treatment groups (EG or CG) and will be clinically and instrumentally evaluated at baseline (T0) and at the end of treatment (T1). EG, in addition to the standard rehabilitation treatment, will perform a 45-minute session of BRAT per day through the Arm Light Exoskeleton Hybrid (Alex RS - Wearable Robotics) robotic system. The CG, in addition to the standard routine rehabilitation treatment, will follow a conventional rehabilitation of the upper limbs without the use of technological devices. Finally, a telephone follow-up is scheduled three months after the end of the treatment.

DETAILED DESCRIPTION:
Cerebral stroke is one of the major causes of mortality and disability in the world. Upper limb disorders are evident up to 85% of stroke survivors and persist, even 6 months after the acute event, in 55-75% of patients. Recovery of upper limb ability represents a major challenge for neurorehabilitation. Among recent strategies and trends in stroke rehabilitation, robotic technologies are having more space and their application in clinical routine is increasing. The promising effects of robot-assisted therapy for upper limb rehabilitation (Robot-Assisted Therapy-RAT) have been demonstrated in terms of recovery of arm and hand range of motion, muscle strength, thus improving performance of activities of daily living (AVQ). In particular, the latest generation exoskeletal robots have demonstrated their effectiveness, promoting a three-dimensional rehabilitation activity. At the same time, bimanual therapy represents a different training modality which has its solid neuroscientific foundations to improve learning and positively address neuroplasticity phenomena. However, there is no information regarding the effectiveness of these robots on subjects suffering from stroke and in the subacute phase. The primary objective of this RCT is to study the clinical effects of upper limb rehabilitation through a bilateral exoskeleton (Bilateral Robot-Assisted Therapy-BRAT) within standard rehabilitation, on motor recovery, compared to conventional arm re-education in people suffering from stroke in the subacute phase. Secondary objectives of the study include: evaluation of the effectiveness of BRAT on bilateral recovery of arm motor skills and quality of life of study participants; the identification of the characteristics of patients who can benefit most from BRAT in terms of age, distance from the acute event and extent of the motor deficit of the upper limb. The effects of BRAT on motor recovery will also be studied from a neurophysiological (EEG and sEMG) and biomechanical (Inertial Measurement Units-IMU) point of view.The study will develop over 24 months, and includes 3 phases as follows: Phase 1- patient enrollment and screening; Phase 2 Treatment of participants; Phase 3 - Statistical analysis of the data. The study protocol will involve people diagnosed with stroke according to established inclusion and exclusion criteria who will be randomly assigned to one of the following groups: Experimental Group (EG) - robotic treatment for upper limb rehabilitation or Control Group (CG) - conventional treatment for upper limb rehabilitation. The experimental group (EG), in addition to the standard rehabilitation treatment, will perform one BRAT session per day through the Arm Light Exoskeleton Hybrid (Alex RS - Wearable Robotics) robotic system. Each participant will perform a total of 16+/-3 treatment sessions with a frequency of 4 times a week for 4 consecutive weeks. All the devices that will be used have the CE (European Conformity) marking. The control group (CG), in addition to the standard routine rehabilitation treatment, will follow a conventional rehabilitation of the upper limbs (16+/-3 treatment sessions) without the use of technological devices. The motor exercises will concern the rehabilitation of the upper limb and will be performed with a therapist who will personalize the treatment based on the clinical characteristics and needs of the patient. Specifically, the treatment of the upper limb will be characterized by motor exercises (shoulder, elbow, wrist and hand), coordination and manual dexterity. All subjects will be evaluated with a standard clinical objective examination and with clinical rating scales and instrumental assessments. These scales will be administered at baseline (T0), at the end of treatment (T1) and 3 months after the end of treatment (follow-up). The main expected results are: identify a customizable rehabilitation protocol for motor recovery of the upper limb based on the clinical characteristics of each individual patient; achieve better motor recovery both in terms of range of motion and muscle recruitment associated with cognitive stimulation following upper limb rehabilitation through the Alex exoskeleton bilateral robotic assistance system; achieve better muscle activation and therefore better motor performance in the EG; achieve greater autonomy in carrying out daily life activities and consequently greater participation.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes;
* Age >18 years;
* Unilateral hemipyramidal syndrome as demonstrated by a brain CT or MRI;
* Distance from acute event < 6 months;
* Modified Ashworth Scale (MAS) of shoulder, elbow, and wrist <3;
* Ability to understand and sign the informed consent for the study;
* Ability to perform the study procedures.

Exclusion Criteria:

* Unstable general clinical conditions;
* Bilateral pyramidal hemisyndrome severe visual impairment;
* Recent injection of Botulinum Toxin to the affected upper limb or planned for the duration of the study;
* Interruption of treatment for 1 week or 5 consecutive sessions;
* Inability to adhere to the exercise program due to poor compliance;
* Presence of neurological pathologies superimposed on the stroke event, psychiatric complications or personality disorders;
* Presence of osteoarticular and neuromuscular pathologies that may compromise the motor skills of the upper limb;
* Participants who have not signed the informed consent to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-05-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Upper Limb Fugle Meyer Assessment - Motor Part (score range: 0-66) | Day 0 (T0- basline) and day 28 (T1 - After treatment)
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. It is applied clinically and in research to determine disease severity, describe motor recovery, and to plan and assess treatment.
  The Fugl-Meyer Assessment (FMA) is a widely used clinical tool to assess motor recovery in individuals who have experienced a stroke. It is designed to measure motor function, sensory function, balance, and joint range of motionin individuals with hemiplegia (one-sided paralysis or weakness), which is common following a stroke.

SECONDARY OUTCOMES:
Oxford Cognitive Scale (OCS) | Day 0 (T0- basline) and day 28 (T1 - After treatment)
  The Oxford Cognitive Screen (OCS) assesses key cognitive domains: memory, language, numerical cognition, praxis, executive functions, and attention. It is designed as a screening tool that enables a rapid evaluation of the patient's cognitive functioning and guides further, more detailed assessment of any impaired cognitive domain(s). It also allows for the evaluation of aphasic patients. Test items are presented both visually and verbally, with the option to select a correct response from multiple choices. To optimize the distribution of attentional resources, the battery items are presented centrally, reducing the need for visual scanning. The OCS allows for the assessment of neglect (both allocentric and egocentric), apraxia, and deficits in numerical cognition.
Modified Ashworth Scale (MAS) 0-4 | Day 0 (T0- basline) and day 28 (T1 - After treatment)
  The Modified Ashworth Scale (MAS) is used to assess spasticity. The Modified Ashworth Scale (MAS) has been utilised in the following populations: stroke, spinal cord injury, multiple sclerosis, cerebral palsy, traumatic brain injury, paediatric hypertonia and central nervous system lesions. The test is performed by extending the patients limb's first from a position of maximal possible flexion to maximal possible extension (the point at which the first soft resistance is met). Afterwards, the modified Ashworth scale is assessed while moving from extension to flexion. Scores range from 0 to 4, where 0 indicates no increase in muscle tone and 4 represents a limb that is rigid in flexion or extension. The score from 0 to 4 indicated in the title refers to the individual joint. Specifically, in this study, the muscle tone of the shoulder, elbow, and wrist will be assessed.
Box and Block test (BBT) | Day 0 (T0- basline) and day 28 (T1 - After treatment)
  The Box and Block Test (BBT) measures unilateral gross manual dexterity. It can be used with a wide range of populations, including clients with stroke.The BBT is composed of a wooden box divided in two compartments by a partition and 150 blocks. The BBT administration consists of asking the client to move, one by one, the maximum number of blocks from one compartment of a box to another of equal size, within 60 seconds.
Nine Hole Peg Test (NHPT) | Day 0 (T0- basline) and day 28 (T1 - After treatment)
  The Nine-Hole Peg Test (9HPT) is used to measure finger dexterity in patients with various neurological diagnoses. The Nine-Hole Peg Test is administered by asking the client to take the pegs from a container, one by one, and place them into holes on the board as quickly as possible. Participants must then remove the pegs from the holes, one by one, and replace them back into the container.Scores are based on the time taken to complete the activity, recorded in seconds.
ABILHAND | Day 0 (T0- basline) and day 28 (T1 - After treatment)
  The ABILHAND is an interview-based assessment of a patient-reported measure of the perceived difficulty in using their hand to perform manual activities in daily activities. The assessment considers the active function of the upper limbs and measures the ability to perform bimanual tasks, regardless of the way in which these tasks are carried out. There are currently versions specifically validated for Chronic stroke, Rheumatoid Arthritis, Systemic sclerosis, Hand Surgery. This is an interview-based assessment where patient is asked to estimate the ease or difficulty of performing a list of activities when carried out without assistance. This can involve any strategy used to carry out the activity, and is self-report and not a physical demonstration of the activity.
  The questionnaire is downloaded from the website and one of the 10 random orders of questions. These are read to the patient and scored as either "impossible", "difficult" or "easy". If a task has not been attempted
Modified Barthel Index (mBI) | Day 0 (T0- basline) and day 28 (T1 - After treatment)
  The modified Barthel Index (mBI) is a well-established patient-centered outcome measure commonly administrated in rehabilitation settings to evaluate the functional status of patients at admission and discharge.
Client Satisfaction Questionnaire (0-24) | Day 28 (T1 - After treatment)
  The Client Satisfaction Questionnaire (CSQ-8) is one of a limited number of standardised satisfaction measures that have been used widely across mental health services.
Frenchay Activities Index (FAI) | Day 120 (T2 - 3 months after treatment Follow-Up)
  The Frenchay Activities Index (FAI) is a measure of instrumental activities of daily living (IADL) for use with patients recovering from stroke. The FAI assesses a broad range of activities associated with everyday life that patient has participated in within the recent past, broken into 3 domains: domestic chores, leisure/work, and outdoor activities. The items included move beyond the scope of ADL scales, which tend to focus on issues related to self care and mobility.
  Can be separated into 3 domains:
  1. Domestic chores
  2. Leisure/work
  3. Outdoor activities The frequency with which each item or activity is undertaken over the past 3-6 months (depending on the nature of the activity) is assigned a score of 1 - 4 where a score of 1 is indicative of the lowest level of activity.
  The scale provides a summed score from 15 - 60.
Disability of the Arm, Shoulder, and Hand (DASH) Questionnarie | Day 120 (T2 - 3 months after treatment Follow-Up)
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is a 30-item questionnaire that looks at the ability of a patient to perform certain upper extremity activities. This questionnaire is a self-report questionnaire that patients can rate difficulty and interference with daily life on a 5 point Likert scale. It has two, 4-item, optional modules used to measure symptoms and function in athletes, artists, and workers who require a high level of function.
  Utilizes a 5-point Likert-Scale measuring from "1" (lowest level of difficulty or severity) to 5" (highest level of difficulty or severity) based on the patient's reported ability to conduct the activities or tasks.
  Total scores range from 0 (minimum) to (100) maximum.

OTHER OUTCOMES:
Instrumental robotic assessment | Day 0 (T0- basline) and day 28 (T1 - After treatment)
  A robotic assessment will be performed only for the subjects in the GS group. The robotic device used in the study allows for the evaluation of: Preliminary measurement of the force exerted by the patient during each movement (isometric contraction); Pre-post measurements of the active Range of Motion (ROM) in the patient's 3D working area and of all the individual joints of the affected arm (constrained joints); Movement precision pre-post (speed peaks recorded during exercises).
Instrumental neurophysiological assessments | Day 0 (T0- basline) and day 28 (T1 - After treatment)
  In a subgroup of GS subjects (neurophysiological pilot study), instrumental assessments of neurophysiological signals will also be performed at centers equipped with the appropriate instruments.
  Surface electromyography (sEMG) and kinematics (stereophotogrammetric system with the RAB protocol) will be recorded during the execution of a standardized motor task (Reaching).
  Electroencephalography (EEG): Brain electrical activity will be recorded from 120 channels during rest conditions with eyes closed and open (5 minutes each). The frequency bands considered will be delta (2-4 Hz), theta (4-8 Hz), Alpha1 (8-10.5 Hz), alpha2 (10.5-13 Hz), beta1 (13-20 Hz), beta2 (20-30 Hz), and gamma (30-40 Hz). The activation current density of cortical sources and brain connectivity will be calculated with the eLORETA software for both hemispheres. Specific networks related to the task performed and the lesioned areas will also be analyzed.
IMU-based targeted Box and Block Test (t-BBT) | Day 0 (T0- basline) and day 28 (T1 - After treatment)
  Instrumental assessment of manual dexterity will be conducted using a sensorized and modified version of the Box and Block Test (BBT). This modified version involves moving 10 cubes from one side of the box to the other positioned on a 5x2 grid. In a subset of EG subjects, kinematic parameters will be measured using Inertial Measurement Units (IMUs), and electrophysiological parameters will be recorded via surface electromyography (sEMG). The assessment will quantify joint kinematics, including range of motion and movement smoothness, as well as upper limb muscle activation patterns, such as muscle onset timing and co-contraction levels. This approach enables a comprehensive evaluation of motor performance during the BBT.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sanaz Pournajaf, DPT, Principal Investigator — IRCCS San Raffaele Roma; Prof. Marco Franceschini, MD, Study Chair — IRCCS San Raffaele Roma
Locations (3):
- Italy (3):
  - San Raffaele Cassino, Cassino, Italy
  - IRCCS San Raffaele Roma, Rome, Italy
  - San Raffaele Sulmona, Sulmona, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared with qualified researchers upon reasonable request, following ethical and regulatory approvals.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Individual participant data (IPD) will be available upon publication of the main results and will remain accessible for at least five years.
Access Criteria: Qualified researchers may request access to the data by submitting a proposal outlining their research objectives. Access will be granted upon ethical and regulatory approval and under a data-sharing agreement.

REFERENCES:
- [Background] Kwakkel G, Kollen BJ, van der Grond J, Prevo AJ. Probability of regaining dexterity in the flaccid upper limb: impact of severity of paresis and time since onset in acute stroke. Stroke. 2003 Sep;34(9):2181-6. doi: 10.1161/01.STR.0000087172.16305.CD. Epub 2003 Aug 7. PMID 12907818
- [Background] Mehrholz J, Pohl M, Platz T, Kugler J, Elsner B. Electromechanical and robot-assisted arm training for improving activities of daily living, arm function, and arm muscle strength after stroke. Cochrane Database Syst Rev. 2018 Sep 3;9(9):CD006876. doi: 10.1002/14651858.CD006876.pub5. PMID 30175845
- [Background] Morone G, Palomba A, Martino Cinnera A, Agostini M, Aprile I, Arienti C, Paci M, Casanova E, Marino D, LA Rosa G, Bressi F, Sterzi S, Gandolfi M, Giansanti D, Perrero L, Battistini A, Miccinilli S, Filoni S, Sicari M, Petrozzino S, Solaro CM, Gargano S, Benanti P, Boldrini P, Bonaiuti D, Castelli E, Draicchio F, Falabella V, Galeri S, Gimigliano F, Grigioni M, Mazzoleni S, Mazzon S, Molteni F, Petrarca M, Picelli A, Posteraro F, Senatore M, Turchetti G, Straudi S; "CICERONE" Italian Consensus Conference on Robotic in Neurorehabilitation. Systematic review of guidelines to identify recommendations for upper limb robotic rehabilitation after stroke. Eur J Phys Rehabil Med. 2021 Apr;57(2):238-245. doi: 10.23736/S1973-9087.21.06625-9. Epub 2021 Jan 25. PMID 33491943
- [Background] Iosa M, Morone G, Ragaglini MR, Fusco A, Paolucci S. Motor strategies and bilateral transfer in sensorimotor learning of patients with subacute stroke and healthy subjects. A randomized controlled trial. Eur J Phys Rehabil Med. 2013 Jun;49(3):291-9. Epub 2012 Nov 20. PMID 23172404
- [Background] Frisoli A, Barsotti M, Sotgiu E, Lamola G, Procopio C, Chisari C. A randomized clinical control study on the efficacy of three-dimensional upper limb robotic exoskeleton training in chronic stroke. J Neuroeng Rehabil. 2022 Feb 4;19(1):14. doi: 10.1186/s12984-022-00991-y. PMID 35120546
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. Int J Surg. 2011;9(8):672-7. doi: 10.1016/j.ijsu.2011.09.004. Epub 2011 Oct 13. No abstract available. PMID 22019563
- [Background] Calabro RS, Naro A, Russo M, Milardi D, Leo A, Filoni S, Trinchera A, Bramanti P. Is two better than one? Muscle vibration plus robotic rehabilitation to improve upper limb spasticity and function: A pilot randomized controlled trial. PLoS One. 2017 Oct 3;12(10):e0185936. doi: 10.1371/journal.pone.0185936. eCollection 2017. PMID 28973024
- [Background] Demeyere N, Riddoch MJ, Slavkova ED, Bickerton WL, Humphreys GW. The Oxford Cognitive Screen (OCS): validation of a stroke-specific short cognitive screening tool. Psychol Assess. 2015 Sep;27(3):883-94. doi: 10.1037/pas0000082. Epub 2015 Mar 2. PMID 25730165
- [Background] Mancuso M, Varalta V, Sardella L, Capitani D, Zoccolotti P, Antonucci G; Italian OCS Group. Italian normative data for a stroke specific cognitive screening tool: the Oxford Cognitive Screen (OCS). Neurol Sci. 2016 Oct;37(10):1713-21. doi: 10.1007/s10072-016-2650-6. Epub 2016 Jul 9. PMID 27395388